CLINICAL TRIAL: NCT04523519
Title: PrEP Intervention for People Who Inject Substances and Use Methamphetamine
Acronym: PRIME
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director of Substance Use Research, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA051850 (NIH); R01DA051850 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video directly observed therapy with contingency management (Experimental): Video directly observed therapy with contingency management, in addition to Integrated Next-Step Counseling.
  Interventions: Behavioral: Video directly observed therapy with contingency management; Behavioral: Integrated Next-Step Counseling
- Integrated Next-Step Counseling (Placebo Comparator)
  Interventions: Behavioral: Integrated Next-Step Counseling

INTERVENTIONS:
Behavioral: Video directly observed therapy with contingency management — PrEP adherence will be assessed by visual recognition software during video capture and reviewed for confirmation by study staff, ensuring that videos demonstrate study medication dosing by participant. Participants will receive small financial incentives upon confirmation of dosing.
  Arms: Video directly observed therapy with contingency management
Behavioral: Integrated Next-Step Counseling — Integrated Next-Step Counseling combines support for behavioral strategies that reduce sexual and injection-related HIV risk and do not involve PrEP, with strategies to support PrEP adherence in brief, client-centered conversations.

SUMMARY:
In this study, "PrEP Intervention for people who Inject Substances and Use Methamphetamine" (PRIME), we propose to assess if using video directly observed therapy with real-time contingency management (VDOT-CM) may help people assigned male sex at birth who inject methamphetamine adhere to PrEP. We will randomize 140 adults who use methamphetamine, are HIV-negative, and have recently engaged in a sexual HIV risk behavior to VDOT-CM or counseling alone for 24 weeks.

The study aims are to (1) determine the efficacy of VDOT-CM compared to counseling alone for PrEP adherence, (2) evaluate the acceptability of PrEP and adherence support strategies among the cohort, and (3) compare injection or chemsex and sexual HIV risk behavior before and during PrEP use.

We hypothesize that participants randomized to VDOT-CM will have superior adherence to PrEP. We also hypothesize that participants will describe barriers to and facilitators of PrEP adherence, and those who are randomized to VDOT-CM will consider it an acceptable PrEP adherence support strategy. Finally, we do not expect to find increased injection, chemsex, or sexual risk behaviors for HIV among study participants after they begin taking PrEP.

DETAILED DESCRIPTION:
New HIV infections among people who inject drugs (PWID) are increasing in the United States and San Francisco. Methamphetamine is a driving force in the transmission of HIV. Multiple studies across diverse populations have found methamphetamine use to be independently associated with both injection and sexual risk behaviors for HIV acquisition. Men who have sex with men (MSM) who inject methamphetamine are at particularly elevated risk for HIV from both injection and sexual risk behaviors.

Daily, oral pre-exposure prophylaxis (PrEP) is safe and highly effective for HIV prevention when taken consistently. The Centers for Disease Control and other health agencies recommend PrEP for PWID. Despite this recommendation and increasing PrEP use in the US, almost no PrEP studies or demonstration projects have focused on PWID. The small number of studies that have evaluated PrEP use among MSM who inject methamphetamine have shown slow PrEP uptake and adherence challenges.

The PRIME study will randomize 140 people assigned male sex at birth who use methamphetamine, are HIV-negative, and have recently engaged in an HIV sexual risk behavior to video directly observed therapy with contingency management (VDOT-CM) and counseling or counseling alone for 24 weeks. The primary aim of this study is to evaluate if VDOT-CM helps people who were assigned male sex at birth who use methamphetamine adhere to daily PrEP for HIV prevention. Participants will be assigned male sex at birth, age 18 years or older, who have used methamphetamine within the past 30 days, are HIV negative and interested in initiating PrEP, and report condomless sero-unknown/discordant sex in the past 12 months. Participants may also be individuals who recently started PrEP with an outside provider.

All subjects will complete the following study visits: screening, enrollment, follow-up visits 6, 12, and 18 weeks from enrollment, and a final follow-up visit at 24 weeks. At screening, enrollment, and all follow-up visits, laboratory testing for HIV, gonorrhea, chlamydia, and methamphetamine metabolites will be done. Syphilis and creatinine testing will be done at screening and week 24. Syphilis testing will also be done at enrollment and week 12. In addition, hepatitis B surface antigen (HBsAg) and hepatitis C antibody (HCV) testing will be done at the screening visit. HCV testing will also be done at the week 24 visit.

At screening a medical history and physical exam will be performed; during enrollment and follow-up a symptom-directed exam will be performed at all visits, and under clinician discretion, a medical history and full exam will be done if needed. AEs will be assessed starting at enrollment and throughout follow-up. Vital signs and weight will be checked at all visits. Some lab procedures will vary if the participant receives PrEP from their own provider or is enrolled remotely.

At enrollment, participants will be randomized 1:1 to receiving only Integrated Next Step Counseling (iNSC) or iNSC and video directly-observed therapy (VDOT) with contingency management (CM). All participants will receive iNSC throughout their participation to support PrEP adherence and help their reduce risk for HIV. Dried blood spots (DBS) will be collected for FTC/TAF drug level testing at weeks 6, 12, 18, and 24. Participants randomized to the VDOT-CM arm will be asked to record taking their daily PrEP dose on VDOT every day from enrollment through week 24.

In-depth interviews will be conducted with at least 36 participants (18/arm) and participants who discontinue PrEP early or become infected with HIV during the study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Age 18-65 years inclusive,
2. Assigned male sex at birth,
3. Past 30-day methamphetamine use on 4 or more days, by self-report,
4. ≥ 1 positive methamphetamine urine toxicology,
5. Either interested in initiating PrEP OR currently on daily PrEP with sub-optimal adherence (measured as missing at least one dose of one's PrEP in the past 30 days, by self-report),
6. Reports condomless sero-unknown/discordant anal or insertive vaginal sex with a person of any gender in the past 12 months,
7. HIV-negative,
8. Reliable access to a computer to complete study visits, if participating remotely, AND
9. Proficient in English

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. On PrEP for more than 6 months,
2. Unwillingness to use a video app to record oneself taking PrEP, OR
3. Any other circumstances that, in the opinion of the investigators, would compromise participant safety and/or successful completion of the trial.

   For participants receiving PrEP from the study team, exclusion criteria will include the following:
4. Contraindication to tenofovir or emtricitabine-containing products,
5. Creatinine clearance ≤30 mL/min, OR
6. Positive hepatitis B surface antigen test.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Tenofovir diphosphate (TFV-DP) levels ≥175 fmol/punch or >= 950 fmol/punch in dried blood spots | Week 6
TFV-DP levels ≥175 fmol/punch or >= 950 fmol/punch in dried blood spots | Week 12
TFV-DP levels ≥175 fmol/punch or >= 950 fmol/punch in dried blood spots | Week 18
TFV-DP levels ≥175 fmol/punch or >= 950 fmol/punch in dried blood spots | Week 24

SECONDARY OUTCOMES:
Qualitative interview data describing participant experiences taking PrEP, with Integrated Next-Step Counseling, and among those randomized to the VDOT-CM arm, experience with VDOT-CM | Interviews done at end of study (24 weeks)
SexPro score | Change in SexPro score from baseline at 12 weeks
  Score that measures sexual HIV risk
SexPro score | Change in SexPro score from baseline at 24 weeks
  Score that measures sexual HIV risk
ARCH-IDU Score | Change in ARCH-IDU score from baseline at 12 weeks
  Score that measures HIV risk related to injection drug use
ARCH-IDU Score | Change in ARCH-IDU score from baseline at 24 weeks
  Score that measures HIV risk related to injection drug use

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Coffin, Principal Investigator — San Francisco Department of Public Health
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Centers for Disease Control and Prevention. HIV Surveillance Report, 2017; vol. 29. http://www.cdc.gov/hiv/library/reports/hiv-surveillance.html. Published 2018. Accessed November 1, 2019
- [Background] San Francisco Department of Public Health. HIV Epidemiology Annual Report 2018. San Francisco Department of Public Health. https://www.sfdph.org/dph/files/reports/RptsHIVAIDS/HIV-Epidemiology-Annual-Report2018.pdf. Published 2019. Accessed November 4, 2019.
- [Background] Degenhardt L, Mathers B, Guarinieri M, Panda S, Phillips B, Strathdee SA, Tyndall M, Wiessing L, Wodak A, Howard J; Reference Group to the United Nations on HIV and injecting drug use. Meth/amphetamine use and associated HIV: Implications for global policy and public health. Int J Drug Policy. 2010 Sep;21(5):347-58. doi: 10.1016/j.drugpo.2009.11.007. Epub 2010 Feb 1. PMID 20117923
- [Background] HIV/AIDS Epidemiology Unit, Public Health - Seattle & King County and the Infectious Disease Assessment Unit, Washington State Department of Health. HIV/AIDS Epidemiology Report & Community Profile 2019, Volume 88.
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Martin M, Vanichseni S, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Curlin ME, Na-Pompet S, Warapronmongkholkul A, Kittimunkong S, Gvetadze RJ, McNicholl JM, Paxton LA, Choopanya K; Bangkok Tenofovir Study Group. The impact of adherence to preexposure prophylaxis on the risk of HIV infection among people who inject drugs. AIDS. 2015 Apr 24;29(7):819-24. doi: 10.1097/QAD.0000000000000613. PMID 25985403
- [Background] Storholm ED, Volk JE, Marcus JL, Silverberg MJ, Satre DD. Risk Perception, Sexual Behaviors, and PrEP Adherence Among Substance-Using Men Who Have Sex with Men: a Qualitative Study. Prev Sci. 2017 Aug;18(6):737-747. doi: 10.1007/s11121-017-0799-8. PMID 28578516
- [Background] Finlayson T, Cha S, Xia M, Trujillo L, Denson D, Prejean J, Kanny D, Wejnert C; National HIV Behavioral Surveillance Study Group. Changes in HIV Preexposure Prophylaxis Awareness and Use Among Men Who Have Sex with Men - 20 Urban Areas, 2014 and 2017. MMWR Morb Mortal Wkly Rep. 2019 Jul 12;68(27):597-603. doi: 10.15585/mmwr.mm6827a1. PMID 31298662
- [Background] Chen YH, Guigayoma J, McFarland W, Snowden JM, Raymond HF. Increases in Pre-exposure Prophylaxis Use and Decreases in Condom Use: Behavioral Patterns Among HIV-Negative San Francisco Men Who have Sex with Men, 2004-2017. AIDS Behav. 2019 Jul;23(7):1841-1845. doi: 10.1007/s10461-018-2299-7. PMID 30306436
- [Derived] McMahan VM, Pope E, Luna Marti X, Walker J, Liu AY, Coffin PO. Interest in Long-Acting Preexposure Prophylaxis (PrEP) Among Men at Risk for Human Immunodeficiency Virus Who Use Methamphetamine Participating in a Daily, Oral PrEP Adherence Trial in San Francisco, California. Open Forum Infect Dis. 2025 May 12;12(5):ofaf280. doi: 10.1093/ofid/ofaf280. eCollection 2025 May. PMID 40406373